CLINICAL TRIAL: NCT03219177
Title: Patient Education and Use of Postoperative Pain Medication in Ambulatory Hand Surgery: a Randomized Controlled Trial
Brief Title: Patient Education and Use of Post Operative Pain Medication in Ambulatory Hand Surgery: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2016-0330
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Ambulatory Hand Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient education group (Experimental)
  Interventions: Behavioral: Patient education regarding indications for opioid use and side effects of opioid use after hand surgery
- Control- Standard of care counseling (Active Comparator)
  Interventions: Other: Standard of care post-operative counseling

INTERVENTIONS:
Behavioral: Patient education regarding indications for opioid use and side effects of opioid use after hand surgery — Patients in the active education group will be given information pre-operatively on the current opioid epidemic, alternative pain management strategies that should be tried before proceeding to prescription opioid use, appropriate indications for opioid use, and side effects of opioids.This information will be reinforced by the research coordinator and nursing staff in the post-anesthesia care unit.
  Arms: Patient education group
Other: Standard of care post-operative counseling — Patients will receive standard of care post-operative counseling. They will not be given pre or post-operative opioid education.
  Arms: Control- Standard of care counseling

SUMMARY:
There is a current opioid epidemic in the United States partially fueled by excess prescribing practices after surgery. The objective of this study is to decrease the amount of opioids needed after ambulatory hand surgery. In this randomized control trial, patients will be randomized into a patient education group and into a control group. The education group will be provided with a pre-operative video detailing proper indications for opioid use after hand surgery, alternative pain management strategies to try before using prescription opioid medications, and side effects associated with opioid use. Patients will also receive information on the current opioid epidemic. Patients will be reminded of the information given pre-operatively after surgery in the post-anesthesia care unit. The control group will not receive pre-operative education and will only receive standard of care post-operative counseling by nursing in the post-anesthesia care unit. All patients will be given a pain log, pain medication diary and participate in phone/email surveys to determine number of opioid pills taken, pain levels, and satisfaction with surgery. The investigators hypothesize that the education group will have decreased opioid intake and increased patient satisfaction compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking: must be able to communicate over the phone or by email to perform questionnaires
* Primary elective ambulatory hand surgery (bony or soft tissue)

Bony: Scaphoidectomy/ligament reconstruction tendon interposition (LRTI), Arthrodesis, Arthroplasty Soft Tissue: Carpal tunnel release (CTR), Trigger Finger (TF), DeQuervain's (DQ), Cyst removal, Cubital tunnel, Dupuytren's, tendon transfer, arthroscopy of wrist or elbow

Exclusion Criteria:

* Disability or preop pain in ipsilateral upper extremity from a secondary condition not related to the study procedure
* Allergy or inability to consume oxycodone, Percocet or Vicodin due to a particular health state
* Current Substance Abuse
* HSS employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Number of prescription opioids used postoperatively | Within 14 days of surgery

SECONDARY OUTCOMES:
Patient satisfaction | Post-op day 3, 8, and 15
  This will be measured on a Likert scale, as used in most orthopedics research.
Pain level | Post-op day 3, 8, 15
  Numeric Rating Scale pain scores
Surgical factors | Recorded on day of surgery
  Type of surgery, length of surgery, type and amount of anesthesia
Pain Catastrophization Score | Measured pre-operatively
  This validated scale is one of the most widely used instruments to evaluate catastrophic thinking related to pain. It specifically evaluates patients' feelings of helplessness and frequency of rumination on and magnification of pain.
Mindfulness Attention Awareness Scale Score | Measured pre-operatively
  This validated scale assesses dispositional mindfulness and has been shown to tap a unique quality of consciousness that is associated with self-regulation and well-being constructs.
Adverse reactions to pain medication | Post-op day 3, 8, 15
  Side effects of opioid and non-opioid medications will be assessed
Prescriptions filled and refilled | Post-op day 3, 8, 15
  We will assess whether patients both initially filled and re-filled their opioid prescriptions
Alternative analgesia used | Post-op day 3, 8, 15
  We will identify if patients use any alternative pain management strategies (i.e., elevation, icing, breathing exercises, mediation, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States